CLINICAL TRIAL: NCT06115668
Title: Effects of Individualized Positive End-Expiratory Pressure (PEEP) on Oxygenation, Hemodynamic Variables, and Incidence of Early Postoperative Atelectasis in Patients Undergoing Laparoscopic Bariatric Surgery: A Prospective Randomized Controlled Study
Brief Title: Individualized Positive End-Expiratory Pressure (PEEP) on Oxygenation, Hemodynamics, and Early Postoperative Atelectasis in Laparoscopic Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Heba Zakaria Mohamed Khattab, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36131/11/22
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Positive End-expiratory Pressure; Hemodynamic Variable; Postoperative Atelectasis; Laparoscopic Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive end-expiratory pressure 5 (PEEP 5) (Active Comparator): Patients will receive fixed positive end-expiratory pressure(= 5 cmH2O) as a control group
  Interventions: Other: Positive end-expiratory pressure 5 (PEEP 5)
- Individualized positive end-expiratory pressure (PEEPIND) (Experimental): Patients who will receive the individualized positive end-expiratory pressure.
  Interventions: Other: Individualized positive end-expiratory pressure (PEEPIND)

INTERVENTIONS:
Other: Positive end-expiratory pressure 5 (PEEP 5) — Fixed positive end-expiratory pressure of 5 cmH2O will be maintained throughout the duration of surgery
  Arms: Positive end-expiratory pressure 5 (PEEP 5)
Other: Individualized positive end-expiratory pressure (PEEPIND) — Patients will receive the individualized positive end-expiratory pressure. Titration process will be started after establishment of pneumoperitoneum: setting the initial PEEP to 5 cmH2O, then increasing positive end-expiratory pressure (PEEP)according to the gradient of 2 cmH2O every 3 min, calculating static compliance (Cstat) according to the formula: [Cstat = VT/Pplat - PEEP] (Pplat = plateau pressure), then gradually increasing positive end-expiratory pressure , until the calculated Cstat shows a downward trend, set its previous PEEP (corresponding to PEEP for high Cstat) as the optimal PEEPIND for this patient. The highest PEEP is limited to 20 cmH2O
  Arms: Individualized positive end-expiratory pressure (PEEPIND)

SUMMARY:
The aim of this study is to evaluate the effectiveness of intraoperative individualized positive end-expiratory pressure (PEEPIND) titration, compared to fixed positive end-expiratory pressure of 5 cmH2O, on oxygenation, hemodynamic variables, and early postoperative complications in obese patients undergoing laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
Obesity is a major health problem, and the incidence is increasing worldwide. So far, the only treatment for morbid obesity with good long-term results is bariatric surgery.

Obese patients have unique respiratory physiology and ventilatory mechanics characteristics. Their lung function is impaired due to the reduction of oxygen reserve, functional residual capacity, and lung compliance. In addition, they frequently present with respiratory comorbidities, which increases the risk of developing postoperative pulmonary complications (PPCs) such as atelectasis especially after procedures under general anesthesia. Atelectasis has been hypothesized as a main cause of postoperative hypoxemia.

To reduce the incidence of atelectasis, positive end-expiratory pressure (PEEP) and recruitment maneuvers are used as a protective lung strategy to improve gas exchange and lung mechanics through reopening collapsed alveoli and maintaining the aeration of lungs. Application of PEEP may also eliminate auto-PEEP without increasing plateau pressure.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 60 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status class I-III
* Patients who are scheduled for elective laparoscopic bariatric surgery under general anesthesia.

Exclusion Criteria:

* Patients who are unwilling to participate in the study
* Actively smokers.
* Patients who had a history of Chronic obstructive pulmonary disease or bronchial asthma.
* Patients who are receiving renal replacement therapy prior to surgery.
* Patients who had a history of heart failure.
* Pregnant.
* Patients who have allergies to any drug used in the study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative oxygenation | One hour after extubation
  Intraoperative oxygenation which will be assessed by P/F ratio (the ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2 expressed as a fraction, not a percentage).
  PaO2/FiO2: will be measured at before induction of anesthesia, immediately after intubation, after PEEP titration, one hour after pneumoperitoneum, before extubation, one hour after extubation

SECONDARY OUTCOMES:
Mean arterial pressure(MAP) | One hour after extubation
  Mean arterial pressure will be measured before induction of anesthesia, immediately after intubation, after positive End-Expiratory Pressure titration, one hour after pneumoperitoneum, before extubation, and one hour after extubation.
Heart rate(HR) | One hour after extubation
  Heart rate will be measured before induction of anesthesia, immediately after intubation, after positive End-Expiratory Pressure titration, one hour after pneumoperitoneum, before extubation, and one hour after extubation.
Volume of total fluid infusion | Till the end of surgery
  The total volume of the administered fluids will be recorded.
Dosage of vasopressors | Till the end of surgery
  The total volume of the administered vasopressors will be recorded.
Lung ultrasound scores | 12 hours postoperatively
  Lung ultrasound scans will be performed 3 times for each patient, before induction of anesthesia, one hour after extubation and 12 hours postoperatively.
  Patients will be scanned in the supine position as follows: Each hemithorax will be divided into 6 regions using 3 longitudinal lines (parasternal, anterior, and posterior axillary) and 2 axial lines (one above the diaphragm and the other 1 cm above the nipples). The 12-lung regions will be scanned sequentially from right to left, cranial to caudal and anterior to posterior. Each region will be assessed using a 2-dimensional view with the probe placed parallel to the ribs. The degree of B-lines will be divided into 4 grades according to lung ultrasound score for consolidation and aeration and scored between 0 and 3:
  (0) fewer than 3 isolated B-lines.
  1. multiple well-defined B-lines.
  2. multiple coalescent B-lines.
  3. white lung.
Early postoperative pulmonary complication | First 24 hours postoperatively
  Any early postoperative pulmonary complication in the first postoperative 24 hours will be recorded.
Length of hospital stay | 28 days postoperatively
  Time from admission till hospital discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.